CLINICAL TRIAL: NCT00573196
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Bipolar Condition
Brief Title: Far Infrared Radiation Treatment for Bipolar Condition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical research Institute Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-BPC-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Bipolar Disorder
Keywords: Affective Psychosis, Bipolar; Depression, Bipolar; Mania; Manic Disorder; Manic State; Manic-Depressive Psychosis; Psychoses, Manic-Depressive; Psychosis, Manic-Depressive
MeSH Terms: conditions — Bipolar Disorder; Mania

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Radiation: Far infrared

INTERVENTIONS:
Radiation: Far infrared — Far infrared radiation (5μm to 15μm wavelength)

SUMMARY:
A preliminary study to determine the possibility of using far infrared radiation for the treatment of the Bipolar Condition

DETAILED DESCRIPTION:
A 2000 study in the American Journal of Psychiatry reported that, "in those with bipolar, two major areas of the brain contain 30 percent more cells that send signals to other brain cells". This fact explains why famous people with the Bipolar condition like astronaut Buzz Aldrin, financier Robert Campeau, British Prime Minister Winston Churchill, composer Mozart, scientist Isaac Newton, physician Sigmund Freud and media giant & entrepreneur Ted Turner, excelled in life due to the additional brain power!

The excessive brain power, however, had to be controlled occasionally with mood stabilizers. Mood stabilizers include a number of anticonvulsants and Lithium. These medications, however, have adverse side effects on the kidneys. The proposed evaluation does not have any adverse health effects.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Bipolar Condition, Depression, Anxiety, Stress and Insomnia

Exclusion Criteria:

* Persons with severe mental illness that are confined to mental hospitals etc. as defined by the USA Diagnostic and Statistical Manual of Mental Disorders (DSM) are excluded from this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on bipolar condition. | 2 years

SECONDARY OUTCOMES:
The secondary end point of the study is to evaluate the therapeutic effects of far infrared radiation on other related mental illness including Depression, Anxiety, Stress and Insomnia. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kwasi Donyina, Ph.D., Principal Investigator — GAAD Medical Research Institute Inc.; Ken Nedd, M.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Mississauga, Ontario, Canada